CLINICAL TRIAL: NCT05047289
Title: Indiana University Gastric Electrical Stimulation Registry
Status: Enrolling by invitation | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Purdue University (Other)
Responsible Party: Principal Investigator, John M. Wo, Director, GI Motility and Neurogastroenterology, Indiana University
Other Study IDs: 2008529997
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Gastroparesis
Keywords: gastroparesis; gastric electrical stimulator; GES; vomiting; nausea; bloating; post prandial fullness; epigastric pain
MeSH Terms: conditions — Gastroparesis; Vomiting; Nausea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

SUMMARY:
The purpose of this study is to develop a clinical registry in patients with Gastric Electrical Stimulation (GES) therapy for gastroparesis to support future gastrointestinal therapies, medical procedures and diagnostics.

DETAILED DESCRIPTION:
This study will evaluate male and female patients at least 18 years of age, with gastroparesis, who will or have already undergone the implantation of a GES device

The study will be conducted at one center and approximately 1,000 subjects will be enrolled.

Subjects undergoing the GES implantation will be enrolled before the implantation and may have a baseline visit. The visit procedures will be conducted at the discretion of the investigator dependent on the clinical condition of the patient at that time.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergo implantation of a new GES device for medical refractory gastroparesis

Exclusion Criteria:

* Non-ambulatory patients: bed-ridden, nursing home resident, etc.
* Pregnancy
* Unable to give own informed consent.
* Prisoners

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will evaluate male and female patients at least 18 years of age, with gastroparesis, who will or have already undergone the implantation of a GES device (Enterra, Medtronic, Minneapolis, MN)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2030-10-20 (Estimated); Study Completion 2030-10-20 (Estimated)

PRIMARY OUTCOMES:
To develop a clinical registry in patients with GES therapy | 3 years
  The purpose of this study is to develop a clinical registry in patients with Gastric Electrical Stimulation (GES) therapy for gastroparesis to support future clinical and translational research. Gastroparesis is an illness caused by a delay of stomach emptying. Symptoms of gastroparesis include nausea, vomiting, weight loss, the feeling of being full right away when you start eating, and abdominal pain. The disease may also lead to malnutrition and weight loss. GES has shown promise in patients with gastroparesis. However, how the GES works is unclear, but the patients who undergo GES show improvement in their symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: John Wo, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States